CLINICAL TRIAL: NCT05198856
Title: A Single-arm, Open, Prospective, Multi-center Study on Thalidomide Combined With First-line Chemotherapy and Monotherapy for Maintenance Treatment of Liver Metastases From Her2-negative Advanced Gastric Cancer
Brief Title: Thalidomide Combined With Chemotherapy and Monotherapy for Maintenance Treatment for Her2-negative Advanced GC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOPE2021-Thal-AGC
Record Dates: First submitted 2021-11-18; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2021-09

CONDITIONS: Gastric Cancer Metastatic to Liver
Keywords: Thalidomide; maintenance treatment; gastric cancer; liver metastases
MeSH Terms: conditions — Stomach Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thalidomide (Experimental): The study is divided into two phases:
  The first phase is a combination phase (chemotherapy +T) : Oxaliplatin (130mg/m2 iv d1) and capecitabine (1000mg/m2 d1-14 po bid) repeated every 21 days for a total of 4-6 cycles. Thalidomide tablet: 100 mg/d, qn, orally.
  The second stage is maintenance stage: Patients who have obtained CR, PR or SD in the first stage enter the maintenance stage and receive maintenance treatment with thalidomide tablets: 100mg/d, qn, orally. Maintained until disease progression or adverse reactions are intolerable.
  Interventions: Drug: Thalidomide Combined With Chemotherapy and Monotherapy

INTERVENTIONS:
Drug: Thalidomide Combined With Chemotherapy and Monotherapy — Combined period：chemotherapy + T ：Thalidomide tablets: 100mg/d
  Maintenance period: 100 mg/d, qn, orally. Sustained to disease progression or intolerable adverse reactions.
  Other Names: Fanyingting

SUMMARY:
The overall incidence of liver metastases from gastric cancer is about 9.9%-18.7%. Gastric cancer has strong heterogeneity and rapid disease progression, and the prognosis of liver metastasis is poor. The 5-year survival rate of patients with liver metastases from gastric cancer is very low, making clinical treatment challenging.

Thalidomide has immunomodulatory and anti-angiogenesis effects. It has been used in the treatment of multiple myeloma for more than 20 years, and there are many clinical studies in solid tumors. In recent years, thalidomide has been found to induce the degradation of IKAROS family transcription factors IKZF1 and IKZF3 in combination with CRBN. Therefore, it is very meaningful to explore the therapeutic value of thalidomide in advanced gastric cancer liver metastasis.

DETAILED DESCRIPTION:
The overall incidence of liver metastases from gastric cancer is about 9.9%-18.7%. Gastric cancer has strong heterogeneity and rapid disease progression, and the prognosis of liver metastasis is poor. The 5-year survival rate of patients with liver metastases from gastric cancer is very low, making clinical treatment challenging. Although immune checkpoint inhibitors have been approved for third-line treatment of advanced gastric cancer, they are expensive and poorly accessible. For patients with poor economic conditions, combination therapy based on chemotherapy regimen or treatment regimen optimization may still be a relatively important direction.

Thalidomide has immunomodulatory and anti-angiogenesis effects. It has been used in the treatment of multiple myeloma for more than 20 years, and there are many clinical studies in solid tumors. In recent years, thalidomide has been found to induce the degradation of IKAROS family transcription factors IKZF1 and IKZF3 in combination with CRBN.

In addition, the sedative effect of thalidomide helps to improve patients' sleep. Thalidomide can also inhibit inflammatory factors such as TNF-α, thus improving appetite and increasing lean body weight in patients with cachexia. Its antiemetic effects can reduce gastrointestinal reactions to chemotherapeutic drugs in combined therapy. Thalidomide is also very cheap in China, which is suitable for patients on long-term maintenance treatment. Therefore, it is of great significance to explore the therapeutic value of thalidomide in liver metastasis of advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years old;
2. ECOG physical status score 0-1 points (within 3 days before starting treatment);
3. Expected survival period ≥ 3 months;
4. Basically normal functions of major organs;
5. Pathologically confirmed metastatic gastric cancer or adenocarcinoma at the gastroesophageal junction with no chance of radical surgery, accompanied by liver metastasis or simple liver metastasis;
6. No previous medical treatment; If neoadjuvant or adjuvant chemotherapy has been performed before and after surgery, recurrence can be defined as first-line therapy only after drug withdrawal for at least six months;
7. HER2 negative. HER2 negative definition: IHC (0 or 1+), or IHC (2+) but negative for FISH (HER2:CEP17<2 with mean HER2 copy number <4.0 signals/cell);
8. Measurable lesions assessed according to RECIST1.1;
9. Able to swallow pills normally.

Exclusion Criteria:

1. Those who are allergic to thalidomide;
2. Pregnant or lactating women;
3. Severe mental illness;
4. Those who cannot take medication or follow up as planned;
5. During the trial period and within 3 months after the trial, the subjects and their partners are not willing to use contraception;
6. Participants in other clinical studies 3 months prior to the trial；
7. Patients who are financially well off and willing to use immune checkpoint inhibitors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2022-03-10 (Estimated); Primary Completion 2024-03-10 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | Randomization to the first occurrence of disease progression or death from any cause up to the clinical cut off date of March10,2024 (up to approximately 18 months) ]
  PFS was defined as the time from randomization to the first occurrence of progressive disease (PD) or death from any cause whichever occurs first as determined by an IRF according to RECIST v1.1. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (including baseline). In addition to the relative increase of 20%, the sum of diameters must also demonstrate an absolute increase of >/= 5 millimeters (mm).

SECONDARY OUTCOMES:
Quality of life (QOL) | UpUp to end of study (up to approximately 24 months)
  EORTC QLQ-C30 (Version 3) Quality of life questionnaire will be used to assess the quality of life of the subjects.
Percentage of Participants With Adverse Events (AEs) | Up to end of study (up to approximately 24 months)
  An adverse event is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Riihimaki M, Hemminki A, Sundquist K, Sundquist J, Hemminki K. Metastatic spread in patients with gastric cancer. Oncotarget. 2016 Aug 9;7(32):52307-52316. doi: 10.18632/oncotarget.10740. PMID 27447571
- [Background] Cheon SH, Rha SY, Jeung HC, Im CK, Kim SH, Kim HR, Ahn JB, Roh JK, Noh SH, Chung HC. Survival benefit of combined curative resection of the stomach (D2 resection) and liver in gastric cancer patients with liver metastases. Ann Oncol. 2008 Jun;19(6):1146-53. doi: 10.1093/annonc/mdn026. Epub 2008 Feb 27. PMID 18304963
- [Background] Xiao Y, Zhang B, Wu Y. Prognostic analysis and liver metastases relevant factors after gastric and hepatic surgical treatment in gastric cancer patients with metachronous liver metastases: a population-based study. Ir J Med Sci. 2019 May;188(2):415-424. doi: 10.1007/s11845-018-1864-4. Epub 2018 Jul 30. PMID 30062399
- [Background] Kang YK, Boku N, Satoh T, Ryu MH, Chao Y, Kato K, Chung HC, Chen JS, Muro K, Kang WK, Yeh KH, Yoshikawa T, Oh SC, Bai LY, Tamura T, Lee KW, Hamamoto Y, Kim JG, Chin K, Oh DY, Minashi K, Cho JY, Tsuda M, Chen LT. Nivolumab in patients with advanced gastric or gastro-oesophageal junction cancer refractory to, or intolerant of, at least two previous chemotherapy regimens (ONO-4538-12, ATTRACTION-2): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2017 Dec 2;390(10111):2461-2471. doi: 10.1016/S0140-6736(17)31827-5. Epub 2017 Oct 6. PMID 28993052
- [Background] Fuchs CS, Doi T, Jang RW, Muro K, Satoh T, Machado M, Sun W, Jalal SI, Shah MA, Metges JP, Garrido M, Golan T, Mandala M, Wainberg ZA, Catenacci DV, Ohtsu A, Shitara K, Geva R, Bleeker J, Ko AH, Ku G, Philip P, Enzinger PC, Bang YJ, Levitan D, Wang J, Rosales M, Dalal RP, Yoon HH. Safety and Efficacy of Pembrolizumab Monotherapy in Patients With Previously Treated Advanced Gastric and Gastroesophageal Junction Cancer: Phase 2 Clinical KEYNOTE-059 Trial. JAMA Oncol. 2018 May 10;4(5):e180013. doi: 10.1001/jamaoncol.2018.0013. Epub 2018 May 10. PMID 29543932
- [Background] Zhou S, Wang F, Hsieh TC, Wu JM, Wu E. Thalidomide-a notorious sedative to a wonder anticancer drug. Curr Med Chem. 2013;20(33):4102-8. doi: 10.2174/09298673113209990198. PMID 23931282
- [Background] Bartlett JB, Dredge K, Dalgleish AG. The evolution of thalidomide and its IMiD derivatives as anticancer agents. Nat Rev Cancer. 2004 Apr;4(4):314-22. doi: 10.1038/nrc1323. No abstract available. PMID 15057291
- [Background] Stewart AK. Medicine. How thalidomide works against cancer. Science. 2014 Jan 17;343(6168):256-7. doi: 10.1126/science.1249543. PMID 24436409
- [Background] Mantovani G, Maccio A, Madeddu C, Serpe R, Massa E, Dessi M, Panzone F, Contu P. Randomized phase III clinical trial of five different arms of treatment in 332 patients with cancer cachexia. Oncologist. 2010;15(2):200-11. doi: 10.1634/theoncologist.2009-0153. Epub 2010 Feb 15. PMID 20156909
- See also: Related Info — http://pubmed.aaaib.top/27447571/
- See also: Related Info — http://pubmed.aaaib.top/18304963/
- See also: Related Info — http://pubmed.aaaib.top/30062399/
- See also: Related Info — http://pubmed.aaaib.top/28993052/
- See also: Related Info — http://pubmed.aaaib.top/29543932/
- See also: Related Info — http://pubmed.aaaib.top/23931282/
- See also: Related Info — http://pubmed.aaaib.top/15057291/
- See also: Related Info — http://pubmed.aaaib.top/24436409/